CLINICAL TRIAL: NCT03789591
Title: Hydroxyurea Optimization Through Precision Study (HOPS): A Prospective, Multi-center, Randomized Trial of Personalized, Pharmacokinetics-guided Dosing of Hydroxyurea Versus Standard Weight-based Dosing for Children With Sickle Cell Anemia.
Brief Title: Hydroxyurea Optimization Through Precision Study
Acronym: HOPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Patrick McGann, Director, Brown University Health Comprehensive Sickle Cell Center, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCHMC_HOPS
Record Dates: First submitted 2018-11-27; First posted 2018-12-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: Hydroxyurea; HbSS; HbSD; TREAT
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is designed with a double-blind design. The clinical provider and participant/family will be aware of the absolute (mg) starting dose and could theoretically calculate the mg/kg starting dose, but the treatment assignment will not explicitly be provided to the provider or the family, and the same procedures will be used for dose escalation or reduction. Although most doses in the Alternative Arm will be different than 20 mg/kg, there are some patients on the standard arm who may have a PK-guided dose that is close to or at 20 mg/kg. Thus, although it may be possible to deduce the study arm, the study is designed technically in a double-blind fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Arm (Active Comparator): Participants randomized to the standard arm will receive a starting dose of hydroxyurea of 20 mg/kg/day.
  Interventions: Drug: Hydroxyurea
- Alternative Arm (Experimental): Participants randomized to the alternative arm will receive a pharmacokinetic guided starting dose of hydroxyurea based on PK labs drawn at a baseline visit to target an area under the curve (AUC) of 115 mg*h/L in an attempt to approximate maximum tolerated dose (MTD). This dose will not exceed the maximum tolerated dose of 35 mg/kg/day.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — The alternative arm will use PK data to choose a starting hydroxyurea dose to achieve an AUC of 115 mg*h/L to approximate maximum tolerated dose. On the standard arm, participants will start at the traditional, weight-based dose of 20 mg/kg/day. Following selection of the starting dose, all participants will follow the same dose escalation and laboratory monitoring procedures.

SUMMARY:
Hydroxyurea Optimization through Precision Study (HOPS) is a prospective, multi-center, randomized trial that will directly compare a novel, individualized dosing strategy of hydroxyurea to standard weight-based dosing for children with SCA. The primary objective of the study is to evaluate whether a pharmacokinetics-based starting hydroxyurea dose thieves superior fetal hemoglobin response to to standard weight-based initial dosing. Patients will be recruited from the pediatric sickle cell clinic at Cincinnati Children's Hospital Medical Center and from additional pediatric sickle cell centers within the United States.

DETAILED DESCRIPTION:
The trial will recruit patients who have decided to initiate hydroxyurea therapy. All participants will have pharmacokinetics studies performed at baseline, following a 20 mg/kg oral dose of hydroxyurea. Pharmacokinetic sampling will use a sparse sampling approach, requiring collection of blood at 3 time points (15 minutes, 60 minutes, 180 minutes) following the hydroxyurea dose. Enrolled participants will be randomized to receive either hydroxyurea using a starting dose of 20 mg/kg/day (Standard Arm) or a personalized PK-guided dose (Alternative Arm) to target an area under the curve (AUC) of 115 mg*h/L based to approximate hydroxyurea exposure seen when patients are escalated to maximum tolerated dose (MTD).

Following randomization and selection of the initial dose, participants in both arms will follow the same procedures of laboratory medication holds for hematological toxicity. The primary endpoint is fetal hemoglobin (HbF) six months following the initiation of hydroxyurea therapy with the hypothesis that participants starting with a PK-guided dose will achieve HbF at least 5% greater than those starting with a 20 mg/kg dose. Based upon the estimated number of new hydroxyurea starts at each site, it is anticipated that it will take 24 months to enroll the 116 participants required to achieve sufficient power to assess the primary endpoint. The study will conclude for each participant 12 months following hydroxyurea initiation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell anemia (HbSS, HbSD, HbS/β0-thalassemia, or similarly severe SCA genotype)
* Age 6 months to 21 years at the time of enrollment
* Clinical decision by patient, family, and healthcare providers to initiate hydroxyurea therapy

Exclusion Criteria:

* Current treatment with chronic, monthly blood transfusions or erythrocytapheresis
* Treatment with hydroxyurea within the past 3 months
* Hemoglobin SC disease, HbS/β+-thalassemia
* Current treatment with other investigational sickle cell medications
* Current known pregnancy or lactation

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Fetal Hemoglobin (HbF) Response Following Six Months of Hydroxyurea Therapy | 6 months after starting daily hydroxyurea therapy
  The primary outcome will be HbF response six months after starting hydroxyurea therapy with the hypothesis that participants in the Alternative Arm (PK-guided starting dose) will have at least 5% higher HbF than the Standard Arm (20 mg/kg starting dose)

SECONDARY OUTCOMES:
F Cells | Baseline, 6 and 12 months after initiating daily hydroxyurea therapy
  In addition to traditional %HbF measurement, F cells will be measured at baseline, 6 months, and 12 months
Gene Expression Patterns of Study Participants | 6 Months after initial Hydroxyurea therapy
  The epigenomic signature and gene expression patterns of study participants receiving hydroxyurea therapy at MTD. MTD is defined as a stable dose without any dose increases (except to account for weight gain), holds, or decreases within 8 weeks with laboratory criteria within the target range. This outcome will explain the mechanisms that yield high HbF responses.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Niss, MD, Principal Investigator — Lifespan
Locations (13):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Hospital of Illinois, Peoria, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Indiana Hemophilia & Thrombosis Center, Inc. (IHTC), Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Cohen Children's Medical Center/Northwell Health, New Hyde Park, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies / University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital., Columbus, Ohio
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Meier ER, Creary SE, Heeney MM, Dong M, Appiah-Kubi AO, Nelson SC, Niss O, Piccone C, Quarmyne MO, Quinn CT, Saving KL, Scott JP, Talati R, Latham TS, Pfeiffer A, Shook LM, Vinks AA, Lane A, McGann PT. Hydroxyurea Optimization through Precision Study (HOPS): study protocol for a randomized, multicenter trial in children with sickle cell anemia. Trials. 2020 Nov 27;21(1):983. doi: 10.1186/s13063-020-04912-z. PMID 33246482